CLINICAL TRIAL: NCT03463330
Title: Benefits of Mild Body Exercises in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00140835
Record Dates: First submitted 2018-03-06; First posted 2018-03-13 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Qigong exercise in intervention arm and mild body exercise in control arm
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participation in the intervention group will involve a total of 14 visits over about 14 weeks to the study site, and then a 6-month follow-up evaluation. Participants will learn and practice the Qigong exercise during the study.
  Interventions: Behavioral: Qigong exercise
- Control Group (Sham Comparator): Participation in the intervention group will involve a total of 14 visits over about 14 weeks to the study site, and then a 6-month follow-up evaluation. Participants will learn and practice a mild body exercise during the study.
  Interventions: Behavioral: Mild body exercise

INTERVENTIONS:
Behavioral: Qigong exercise — The Qigong exercise is a series of mild exercise movements.
  Arms: Intervention Group
Behavioral: Mild body exercise — Participants will be taught of series of similar movements to the Qigong exercise.
  Arms: Control Group

SUMMARY:
The purpose of this study is to learn the effects of two mild body exercises on quality of life, non-motor symptoms, anxiety, depression, fatigue, sleep quality, cognition, and executive function on people with Parkinson's Disease (PD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD
* Currently taking levodopa with some improvement in motor symptoms, and on a stable dose for a minimum of 4 weeks prior to starting the study
* Hoehn & Yahr stage I to III (mild to moderate PD)

Exclusion Criteria:

* Mini Mental State Examination (MMSE) score < 24
* Central neurological diseases other than PD or prior major head trauma with loss of consciousness, including other forms of parkinsonism, uncontrolled or significant cardiovascular diseases, orthopedic or medical problems that would interfere with gait
* Being primarily wheelchair bound
* Deep brain stimulation
* Expected change in PD medications over the course of the study
* Subjects with MRI contraindications such as pacemaker, aneurysm clips, artificial heart valves, metal fragments, foreign objects or claustrophobia.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Parkinson's Disease Sleep Scale (PDSS-2) | Change from Baseline to Week 12
  This instrument has a total range of scores between 0 and 60. The lower the score the better.

SECONDARY OUTCOMES:
Parkinson's Disease Questionnaire (PDQ-39) | Change from Baseline to Week 12
  Measure of quality of life. This instrument has a total range of scores between 0 and 156. The lower the score the better.
Non Motor Symptom Questionnaire (NMSQuest) | Change from Baseline to Week 12
  This instrument has a total range of scores between 0 and 30. The lower the score the better.
Geriatric Anxiety Scale (GAS-10) | Change from Baseline to Week 12
  This instrument has a total range of scores between 0 and 30. The lower the score the better.
Geriatric Depression Scale (GDS-15) | Change from Baseline to Week 12
  This instrument has a total range of scores between 0 and 15. The lower the score the better.
Parkinson Fatigue Scale (PFS-16) | Change from Baseline to Week 12
  This instrument has a total range of scores between 16 and 90. The lower the score the better.
Parkinson's Disease-Cognitive Rating Scale (PD-CRS) | Change from Baseline to Week 12
  This instrument has a total range of scores between 0 and 134. The higher the score the better.
Frontal Assessment Battery (FAB-18) | Change from Baseline to Week 12
  This instrument has a total range of scores between 0 and 18. The higher the score the better.
Trail Making Test parts A | Change from Baseline to Week 12
  This test examines the time required to complete a task of connecting numbers in ascending sequence.
Trail Making Test parts B | Change from Baseline to Week 12
  This test examines the required time for completing a task of connecting numbers and letters in ascending sequence.
Unified Parkinson Disease Rating Scale (UPDRS) | Change from Baseline to Week 12
  This instrument has a total range of scores between 0 and 199. The lower the score the better.
IL-1beta | Change from Baseline to Week 12
  Serum biomarker will be measured by Enzyme Linked Immuno-Sorbent Assay (ELISA).
IL-6 | Change from Baseline to Week 12
  Serum biomarker will be measured by Enzyme Linked Immuno-Sorbent Assay (ELISA).
TNF-alpha | Change from Baseline to Week 12
  Serum biomarker will be measured by Enzyme Linked Immuno-Sorbent Assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Wen Liu, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share all IPD data that underlie results in our publications.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The shared information will be available in our lab webpage 6 months after publication.
Access Criteria: The data will be shared with researchers who plan to conduct meta analysis. The PI will review any request for data sharing and make decisions on data sharing.
URL: https://www.kumc.edu/school-of-health-professions/academics/departments/physical-therapy-rehabilitation-science-and-athletic-training/research/neuromuscular-research-laboratory.html

REFERENCES:
- [Background] Moon S, Sarmento CVM, Colgrove Y, Liu W. Complementary Health Approaches for People With Parkinson Disease. Arch Phys Med Rehabil. 2020 Aug;101(8):1475-1477. doi: 10.1016/j.apmr.2020.03.024. Epub 2020 Jul 3. No abstract available. PMID 32631594
- [Background] Moon S, Sarmento CVM, Smirnova IV, Colgrove Y, Lyons KE, Lai SM, Liu W. Effects of Qigong Exercise on Non-Motor Symptoms and Inflammatory Status in Parkinson's Disease: A Protocol for a Randomized Controlled Trial. Medicines (Basel). 2019 Jan 18;6(1):13. doi: 10.3390/medicines6010013. PMID 30669324
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- See also: The shared IPD will be accessible to researchers on our lab webpage. — https://www.kumc.edu/school-of-health-professions/academics/departments/physical-therapy-rehabilitation-science-and-athletic-training/research/neuromuscular-research-laboratory.html